CLINICAL TRIAL: NCT04116086
Title: Using PSMA PET-CT as a Diagnostic Tool for Detection of Prostatic Cancer at an Early Stage
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Dr. Tima Davidson, Head of the Hybrid Imaging Unit, Sheba Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SHEBA-19-6243-TD-CTIL
Record Dates: First submitted 2019-09-11; First posted 2019-10-04 (Actual); Last update posted 2019-10-04 (Actual); Status verified 2019-10

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: One investigator will interpret the PSMA PET-CT and another one will interpret MRI, both in a blinded and independent fashion and before the biopsy. At the end of the study, these 'blind' PSMA PET-CT and MRI reports will be compared to each other and to the actual fusion biopsy results. In the event that a high correlation is found between the diagnostic imaging results to those of the fusion biopsies, it would suggest that PSMA PET-CT could give the option to be performed instead of the need for biopsy in men who present with high levels of PSA and prompt treatment accordingly.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PSMA PET-CT exam (Other): Ga 68 -PSMA PET/CT scanning will be performed using a combined PET/CT protocol with a 16-detector-row helical CT scanner (Philips Gemini GXL). This scanner allows simultaneous acquisition of up to 45 transaxial PET images with interslice spacing of 5 mm in one bed position and provides an image from the vertex to the thigh in about 10 bed positions. The use of (68)Ga-PSMA HBED-CC results in a relatively low radiation exposure, delivering organ doses that are comparable to those of other (68)Ga-labelled PSMA-inhibitors used for PET-imaging. Total effective dose is lower than for other PET-agents used for prostate cancer imaging (e.g. (11) C- and (18) F-Choline).
  Interventions: Diagnostic Test: Prostate Biopsy Test

INTERVENTIONS:
Diagnostic Test: Prostate Biopsy Test — see earlier information
  Other Names: PSMA PET-CT Imaging

SUMMARY:
The aim of the study is the evaluation of the possible role of PSMA PET-CT in early detection of prostate cancer, reducing rate of unnecessary prostate biopsies, and in cases of prostate cancer, correct staging of the disease and corresponding management.

DETAILED DESCRIPTION:
The aim of the study is the evaluation of the possible role of PSMA PET-CT in early detection of prostate cancer, reducing rate of unnecessary prostate biopsies, and in cases of prostate cancer, correct staging of the disease and corresponding management.

Consequently, use of PSMA PET-CT in patients with suspicious PSA changes may improve our knowledge whether the prostate tumor is clinically significant or not (for the development of PSMA PET-CT with 68 Ga ligand allows to visualize prostate cancer with aggressive patterns), and improve clinical decision making for performing prostate biopsy or selecting patients for observation only.

In light of the above, we are of the opinion that this proposed study has the potential to significantly alter the medical practice of how prostate cancer is diagnosed, which even today suffers from real clinical dilemma.

ELIGIBILITY:
Inclusion Criteria:

1. Men aged 40-75
2. With or without suspicious DRE,
3. Were referred by their treating physicians for prostate cancer biopsy based on either an elevated PSA result, a suspicious DRE exam, or both
4. 4 < PSA ≤ 10 ng/ml

   -

   Exclusion Criteria:
5. A previous diagnosis of prostate cancer
6. Underwent previous prostate biopsy
7. Previous radiation to pelvis for any reason

   -

Ages: 40 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 50 (Estimated)
Dates: Start 2019-09-11 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Prostate Cancer Diagnosis | 2 months
  One investigator will interpret the PSMA PET-CT and another one will interpret MRI, both in a blinded and independent fashion and before the biopsy. At the end of the study, these 'blind' PSMA PET-CT and MRI reports will be compared to each other and to the actual fusion biopsy results. In the event that a high correlation is found between the diagnostic imaging results to those of the fusion biopsies, it would suggest that PSMA PET-CT could give the option to be performed instead of the need for biopsy in men who present with high levels of PSA and prompt treatment accordingly.

CONTACTS AND LOCATIONS:
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel

IPD SHARING:
Plan to Share IPD: No